CLINICAL TRIAL: NCT00333736
Title: Prospective Study to Assess Patient Satisfaction, Quality of Life and Adverse Events of Patients Using the Biojector Versus Standard Needles for Enfuvirtide Administration
Brief Title: Study to Assess Safety and Quality of Life of Patients Using Biojector Versus Needles for Fuzeon Administration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Immunodeficiency Research Collaborative (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Roche-B1.0
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Human Immunodeficiency Virus
Keywords: Injection site reactions; enfuvirtide administration
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Injection Site Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Biojector — All patients received biojector to use with BID enfuvirtide doses

SUMMARY:
Hypothesis: Patients using enfuvirtide with the Biojector have an improved quality of life, greater satisfaction, and fewer adverse events compared with using the standard needle.

DETAILED DESCRIPTION:
This study is a "N of one" trial where the patient is their own control. We will provide the quality of life questionnaire, the MOS-HIV questionnaire; ISR questionnaire and a satisfaction questionnaire to patients that have used a standard need to inject enfuvirtide for at least one month. As well, demographics and laboratory data will be collected. The same procedures will be given 1 month after the use of Biojector in a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

Patients who have taken enfuvirtide for at least one month

Exclusion Criteria:

Patients with hemophilia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 337 (Actual)
Dates: Start 2005-05; Primary Completion 2007-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To compare quality of life, satisfaction, and adverse events in patients using a Biojector® versus using a standard needle system for administration of enfuvirtide. | 1 month
  To compare quality of life, satisfaction, and adverse events in patients using a Biojector® versus using a standard needle system for administration of enfuvirtide.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Loutfy, MD, FRCP(C), Principal Investigator — University of Toronto
Locations (1):
- Maple Leaf Medical Clinic, Toronto, Ontario, Canada